## Comparison of the Effectiveness of USG and Palpation Guidance Steroid Injection in Patients With Plantar Fasciitis

## NCT04709484 - 01.03.2021

66 (sixty-six) patients were included in the study. Patients diagnosed with plantar fasciitis, aged between 18-75 years, with failure of conservative treatment (stretching exercises, non-steroidal anti-inflammatory drugs and heel pads) for at least 3 months, with a Visual Analogue Scale value of 5 and above were included in the study. Receiving any local injection therapy and physical therapy for heel pain in the last 4 months, any history of surgery for heel pain, history of tarsal tunnel syndrome, ankle effusion showing intra-articular disease, old healed calcaneal fracture, Achilles tendinopathy, foot and foot any wrist deformity, planus or pes cavus deformity; Patients with systemic disorders such as diabetes mellitus, rheumatoid arthritis, hematological disease or gout, pregnancy, recent history of aspirin or aspirin-like medication, and mental disability were excluded from the study.

In the study, patients' Visual Analogue Scale (VAS) and Foot Function Index (FFI) questionnaires were filled. Patients were randomized into 2 groups according to Random Number Generation. The first group was designed as the USG guided steroid injection group, and the second group was designed as the palpation guided steroid injection group. 34 patients were included in the 1st group and 32 patients in the 2nd group. The patients in the USG group were injected with steroids to the thickened area of the fascia under USG guidance. In the palpation guided practice, the most painful point was found by palpation of the calcaneus bone and steroid injection was made to that part. The content of the steroid solution was 1 ml of 1% Lidocaine + 1 ml (40 mg) of methylprednisolone. There will be pre-injection, post-injection 1st and 3rd month controls.